CLINICAL TRIAL: NCT00000814
Title: A Comparative Study of Combination Antiretroviral Therapy in Children and Adolescents With Advanced HIV Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: ACTG 245; 11222 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-10-28 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: Didanosine; Drug Therapy, Combination; Acquired Immunodeficiency Syndrome; AIDS-Related Complex; Zidovudine; Nevirapine
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome; AIDS-Related Complex | interventions — Nevirapine; Zidovudine; Didanosine

INTERVENTIONS:
Drug: Nevirapine
Drug: Zidovudine
Drug: Didanosine

SUMMARY:
To compare the antiviral activity, safety, toxicity, and steady-state pharmacokinetics of zidovudine, didanosine, and nevirapine used in combination in patients with HIV infection.

The duration of clinical benefit from zidovudine (AZT) may be limited because of development of viral resistance to the drug. Use of combination antiretroviral therapy can potentially reduce viral load and prevent emergence of multidrug resistance.

DETAILED DESCRIPTION:
The duration of clinical benefit from zidovudine (AZT) may be limited because of development of viral resistance to the drug. Use of combination antiretroviral therapy can potentially reduce viral load and prevent emergence of multidrug resistance.

In Stage 1 of the study, a minimum of 22 patients are randomized to each of three treatment arms: didanosine (ddI) plus AZT plus nevirapine (NVP); ddI plus AZT; and ddI plus NVP. After 12 weeks of treatment, the study proceeds to Stage 2 provided at least 40 percent of patients in Stage 1 show a reduction of at least 40 percent from baseline ICD p24 antigen of greater than or equal to 70 pg/ml AND fewer than two patients experience grade 4 rash. Patients in Stage 1 continue treatment for an additional 36 weeks. In Stage 2, additional patients are randomized to each original treatment regimen until a maximum of 130 patients per arm have been entered. Stage 2 patients receive treatment for at least 48 weeks.

AS PER AMENDMENT 02/12/97: As of 2/28/97, patients receiving study drugs will be offered blinded study drugs for an additional 16 weeks (until 6/30/97). Patients will be unblinded on or about 5/23/97.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Erythropoietin.

Concurrent Treatment:

Allowed:

* Transfusion.

Patients must have:

* Progressive HIV disease.
* At least 24 weeks prior cumulative nucleoside analog antiretroviral monotherapy or combination therapy.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

* Active malignancy requiring chemotherapy.
* Currently receiving therapy in an ACTG primary therapy or salvage protocol who have NOT met an endpoint on that study.
* Known intolerance (other than hematologic) or toxicity to ddI, AZT, or NVP at the doses used in this study.

Concurrent Medication:

Excluded (unless exemption made by study chair):

* Oral anticoagulants (warfarin, dicumarol).
* Oral contraceptives.
* Digitalis glycosides.
* Phenytoin.
* Theophylline.

Patients with the following prior conditions are excluded:

* History of clinical pancreatitis.
* History of grade 2 or worse peripheral neuropathy.

Prior Treatment:

Excluded:

* Acute treatment for a serious bacterial, viral, or opportunistic infection within 14 days prior to study entry.

Ages: 6 Months to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 390
Dates: Study Completion 1998-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Burchett S, Study Chair; Luzuriaga K, Study Chair
Locations (68):
- United States (65):
  - Univ of Alabama at Birmingham Schl of Med / Pediatrics, Birmingham, Alabama
  - UCSD Med Ctr / Pediatrics / Clinical Sciences, La Jolla, California
  - Long Beach Memorial (Pediatric), Long Beach, California
  - Los Angeles County - USC Med Ctr, Los Angeles, California
  - Cedars Sinai / UCLA Med Ctr, Los Angeles, California
  - UCLA Med Ctr / Pediatric, Los Angeles, California
  - Harbor - UCLA Med Ctr / UCLA School of Medicine, Los Angeles, California
  - Children's Hosp of Oakland, Oakland, California
  - UCSF / Moffitt Hosp - Pediatric, San Francisco, California
  - Children's Hosp of Denver, Denver, Colorado
  - Univ of Connecticut / Farmington, Farmington, Connecticut
  - Yale Univ Med School, New Haven, Connecticut
  - Georgetown Univ Med Ctr, Washington D.C., District of Columbia
  - Children's Hosp of Washington DC, Washington D.C., District of Columbia
  - Howard Univ Hosp, Washington D.C., District of Columbia
  - Univ of Florida Health Science Ctr / Pediatrics, Jacksonville, Florida
  - Univ of Miami (Pediatric), Miami, Florida
  - Emory Univ Hosp / Pediatrics, Atlanta, Georgia
  - Cook County Hosp, Chicago, Illinois
  - Univ of Illinois College of Medicine / Pediatrics, Chicago, Illinois
  - Chicago Children's Memorial Hosp, Chicago, Illinois
  - Univ of Chicago Children's Hosp, Chicago, Illinois
  - Tulane Univ / Charity Hosp of New Orleans, New Orleans, Louisiana
  - Univ of Maryland at Baltimore / Univ Med Ctr, Baltimore, Maryland
  - Johns Hopkins Hosp - Pediatric, Baltimore, Maryland
  - Children's Hosp of Boston, Boston, Massachusetts
  - Baystate Med Ctr of Springfield, Springfield, Massachusetts
  - Univ of Massachusetts Med School, Worcester, Massachusetts
  - Children's Hosp of Michigan, Detroit, Michigan
  - UMDNJ - Robert Wood Johnson Med School / Pediatrics, New Brunswick, New Jersey
  - Saint Joseph's Hosp and Med Ctr/UMDNJ - New Jersey Med Schl, Newark, New Jersey
  - Children's Hosp at Albany Med Ctr, Albany, New York
  - King's County Hosp Ctr / Pediatrics, Brooklyn, New York
  - SUNY - Brooklyn, Brooklyn, New York
  - North Shore Univ Hosp, Great Neck, New York
  - Schneider Children's Hosp, New Hyde Park, New York
  - Beth Israel Med Ctr / Pediatrics, New York, New York
  - Bellevue Hosp / New York Univ Med Ctr, New York, New York
  - Cornell Univ Med College, New York, New York
  - Metropolitan Hosp Ctr, New York, New York
  - Mount Sinai Med Ctr / Hemophilia Treatment Ctr, New York, New York
  - Mount Sinai Med Ctr / Pediatrics, New York, New York
  - Columbia Presbyterian Med Ctr, New York, New York
  - Incarnation Children's Ctr / Columbia Presbyterian Med Ctr, New York, New York
  - Harlem Hosp Ctr, New York, New York
  - Univ of Rochester Medical Center, Rochester, New York
  - State Univ of New York at Stony Brook, Stony Brook, New York
  - SUNY Health Sciences Ctr at Syracuse / Pediatrics, Syracuse, New York
  - Bronx Lebanon Hosp Ctr, The Bronx, New York
  - Bronx Municipal Hosp Ctr / Bronx Lebanon Hosp Ctr, The Bronx, New York
  - Westchester Hosp, Valhalla, New York
  - Duke Univ Med Ctr, Durham, North Carolina
  - Univ of North Carolina at Chapel Hill / Duke Univ Med Ctr, Durham, North Carolina
  - Columbus Children's Hosp, Columbus, Ohio
  - West Central Ohio Hemophilia Ctr / Children's Med Ctr, Dayton, Ohio
  - Milton S Hershey Med Ctr, Hershey, Pennsylvania
  - Univ of Pittsburgh Med School / Hershey Med Ctr, Hershey, Pennsylvania
  - Children's Hosp of Philadelphia, Philadelphia, Pennsylvania
  - Saint Christopher's Hosp for Children, Philadelphia, Pennsylvania
  - Rhode Island Hosp / Brown Univ, Providence, Rhode Island
  - Med Univ of South Carolina, Charleston, South Carolina
  - Children's Med Ctr of Dallas, Dallas, Texas
  - Texas Children's Hosp / Baylor Univ, Houston, Texas
  - Children's Hosp of the King's Daughters, Norfolk, Virginia
  - Children's Hospital & Medical Center / Seattle ACTU, Seattle, Washington
- Puerto Rico (3):
  - Ramon Ruiz Arnau Univ Hosp / Pediatrics, Bayamón
  - Univ of Puerto Rico / Univ Children's Hosp AIDS, San Juan
  - San Juan City Hosp, San Juan

REFERENCES:
- [Background] McKinney RE Jr. Ongoing and future trials of antiretroviral therapy in the pediatric AIDS clinical trials group (PACTG). Conf Retroviruses Opportunistic Infect. 1996 Jan 28-Feb 1;3rd:173
- [Background] Burchett SK, Carey V, Yong F, Sullivan J, Sulzbacher S, Civitello L, Culnane M, Mofenson L, Siminski S, Robinson P, Luzuriaga K. Virologic activity of didanosine (ddI), zidovudine (ZDV) and nevirapine (NVP) combinations in pediatric subjects with advanced HIV disease (ACTG 245). Conf Retroviruses Opportunistic Infect. 1998 Feb 1-5;5th:130 (abstract no 271)
- [Background] Perrier M, Schwarz T, Gonzalez O, Brounts S. Squamous cell carcinoma invading the right temporomandibular joint in a Belgian mare. Can Vet J. 2010 Aug;51(8):885-7. PMID 21037891
- [Background] Burchett S, Sullivan J, Luzuriaga K, Carey V, Yong F, Culnane M, Mofenson L, Robinson P. Combinations of didanosine (DDI), zidovudine (ZDV) and nevirapine (NVP) can reduce CSF HIV-1 viral load in pediatric patients with advanced HIV disease. Int Conf AIDS. 1998;12:62 (abstract no 12253)